CLINICAL TRIAL: NCT05937256
Title: Quadratus Lumborum Block Versus Erector Spinae Plane Block As Analgesic Alternatives During Extracorporeal Shock Wave Lithotripsy
Brief Title: Quadratus Lumborum Block Versus Erector Spinae Plane Block in Extracorporeal Shock Wave Lithotripsy(ESWL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Gaber Ahmed, Lecturer in anesthesiology, intensive care and pain management, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Regional blocks in ESWL
Record Dates: First submitted 2023-05-28; First posted 2023-07-10 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Pain; Lithiasis
MeSH Terms: conditions — Pain; Lithiasis

STUDY DESIGN:
Intervention Model Description: controlled, randomized, assessor blinded clinical trial.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group Q (Active Comparator): (n=30) will receive unilateral quadratus lumborum block type III
  Interventions: Procedure: Quadratus lumborum block type III
- Group E (Active Comparator): (n=30) will receive unilateral erector spinae plane block
  Interventions: Procedure: Erector spinae plane block
- Group C (No Intervention): (n=30) will be control group receiving no intervention, managed only with conventional analgesia

INTERVENTIONS:
Procedure: Quadratus lumborum block type III — Patients will be placed in lateral decubitus position with the side of the target stone facing up. After sterilization and draping of the skin, using US probe the block will be applied targeting the fascial plane between the quadratus lumborum and psoas major muscles (anterior aspect of the quadratus lumborum). After 20 min, sensory blockade will be evaluated with pinprick test, if loss of sensation is achieved at the T7-L1 dermatome site, the block is considered successful and patients will be transferred to ESWL Room.
  Arms: Group Q
Procedure: Erector spinae plane block — Patients will be placed in the lateral decubitus position according to the selected site. After sterilization and draping of the skin, using US probe, the block will be applied in the plane deep to the erector spinae muscles and superficial to the transverse process. After 20 min, sensory blockade will be assessed with pinprick test, if loss of sensation is achieved at the T7-L1 dermatome site, the block is considered successful and patients is transferred to ESWL Room.
  Arms: Group E

SUMMARY:
This study is designed to compare analgesic effect of both the ultrasound (US)-guided QLB and ESPB blocks during ESWL and their effect on stone fragmentation.

DETAILED DESCRIPTION:
Urinary tract calculi, one of the most common benign urological diseases, is seen in 12% of patients and has a recurrence rate of approximately 50%.

Management of renal calculi is known to be affected by many factors, specially tolerance of pain during ESWL and how it is controlled.

Pain experienced during ESWL is thought to occur when shock waves from the lithotripter reach superficial structures such as skin and also deeper structures such as the ribs, nerves and the kidney capsule. There are three main factors that contribute to the propagation of pain at these structures: shock wave (SW) pressure, distribution, and focal area size .

Conventionally, pain during ESWL is managed by basic analgesics such as NSAIDs, which can also aid in stone clearance. Other methods of analgesia also have been studied and tested.

Quadratus lumborum block (QLB) was first described by Blanco in 2007, it blocks T7-L1 nerve fibres in most of the cases. Studies have reported its use in the management of postoperative pain after hip surgeries.

"Erector Spinae Plane Block" (ESPB) is another such block, that is increasingly tried for the management of postoperative pain for breast surgery, thoracic surgery, and also upper abdominal surgeries. ESPB when given at the lumbar region gives blockade from C7-T2 to L2-L3.

ELIGIBILITY:
Inclusion Criteria:

* Informed written consent obtained
* Age 18-60
* Both sex
* American Society of Anesthesiologists(ASA) physical status: I, II
* Stone pelvis less than 2.5 cm
* Indicated for ESWL

Exclusion Criteria:

* refusal of participation by parents or caregivers.
* ASA physical status: > II
* Stone pelvis >2.5 cm
* Chronic pain
* On chronic NSAID or opioid
* Substance addict
* Known local anesthetic drug sensitivity.
* Preexisting infection at block site
* Coagulopathy or anticoagulation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Analgesic Effect: cumulative opioid dose | At 30 minutes
  Comparing analgesic Effect of both QLB and ESPB by calculating the total opioid consumption over the total duration of session (approximately 30 minutes)

SECONDARY OUTCOMES:
Stone fragmentation: clearance rate | one week after ESWL session
  Determining if stone fragmentation considered satisfactory or not, by Follow up kidney, ureter and bladder x-ray (KUB) and Ultrasound.
Stone fragmentation: shockwave energy | at 30 minutes
  the level of energy will increase gradually, with shock waves between 3,500 and 5,000 in the 2-4 kilovolt (kV) energy range. Fluoroscopy will be used to check the stone and confirm fragmentation. Then maximum and mean energy of shock that is used will be calculated at the end of session approximately 30 min
Block failure rate | Immediately After 20 minutes of intervention
  the block will be considered a failed block if the sensory block level of T7-L1 is not achieved after assessment with pinprick test.
The regional block time | procedure (At the end of intervention)
  defined as the time taken from the start of the ultrasound scan to the completion of the local anesthetic injection.
Feasibility of visualisation | procedure (At the end of intervention)
  The ultrasound images will be evaluated with a 4-point method(10) : 0 points, unable to display; 1 point, the anatomical structure and injection target position are not clear, and the puncture needle is partially developed; 2 points, the anatomical structure, and injection target position are clear, but the puncture needle tip is poorly developed, and local anesthetic diffusion is limited; 3 points, typical anatomical structure, and injection target position, the puncture needle tip can be accurately identified, and local anesthetic diffusion is complete. Images with ≥2 points meant that local anesthetics could be injected.
Adverse effects | immediately after 20 minutes of intervention
  The incidence of adverse effects local (anesthetic toxic reactions, bleeding, or hematoma at the puncture position; failure of block).
Patient satisfaction | At 30 minutes
  patient satisfaction will be recorded after the procedure using a five-point scale, where 1 is unsatisfied and 5 completely satisfied. At the end of session approximately 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed G Ahmed, MD, Principal Investigator — Lecturer in anesthesiology intensive care and pain management, South Valley University
Locations (1):
- South Valley University, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yayik AM, Ahiskalioglu A, Alici HA, Celik EC, Cesur S, Ahiskalioglu EO, Demirdogen SO, Karaca O, Adanur S. Less painful ESWL with ultrasound-guided quadratus lumborum block: a prospective randomized controlled study. Scand J Urol. 2019 Dec;53(6):411-416. doi: 10.1080/21681805.2019.1658636. Epub 2019 Sep 9. PMID 31496381
- [Background] Yayik AM, Celik EC, Ahiskalioglu A. An unusual usage for ultrasound guided Quadratus Lumborum Block: Pediatric extracorporeal shock wave lithotripsy. J Clin Anesth. 2018 May;46:47-48. doi: 10.1016/j.jclinane.2018.01.016. Epub 2018 Mar 26. No abstract available. PMID 29414615
- [Background] Bovelander E, Weltings S, Rad M, van Kampen P, Pelger RCM, Roshani H. The Influence of Pain on the Outcome of Extracorporeal Shockwave Lithotripsy. Curr Urol. 2019 Mar 8;12(2):81-87. doi: 10.1159/000489424. PMID 31114465
- [Background] Oh SK, Lim BG, Won YJ, Lee DK, Kim SS. Analgesic efficacy of erector spinae plane block in lumbar spine surgery: A systematic review and meta-analysis. J Clin Anesth. 2022 Jun;78:110647. doi: 10.1016/j.jclinane.2022.110647. Epub 2022 Jan 11. PMID 35030493
- [Background] El-Boghdadly K, Desai N, Halpern S, Blake L, Odor PM, Bampoe S, Carvalho B, Sultan P. Quadratus lumborum block vs. transversus abdominis plane block for caesarean delivery: a systematic review and network meta-analysis. Anaesthesia. 2021 Mar;76(3):393-403. doi: 10.1111/anae.15160. Epub 2020 Jul 4. PMID 32621529